CLINICAL TRIAL: NCT03069183
Title: The Efficacy of Ultrasound-guided Suprainguinal Fascia Iliaca Compartment Block on Early Post-operative Analgesia After Total Hip Arthroplasty
Brief Title: Ultrasound-guided Suprainguinal Fascia Iliaca Compartment Block for Analgesia After Total Hip Arthroplasty
Acronym: HIPFIB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 838-2017
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2018-07

CONDITIONS: Arthritis of Hip
Keywords: Fascia Iliaca Block; Total Hip Arthroplasty; Total Hip Replacement; Ultrasound
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.5% Ropivacaine (Active Comparator): Ultrasound-guided suprainguinal fascia iliaca compartment block with 40mls 0.5% ropivacaine.
  Interventions: Drug: 0.5% Ropivacaine
- Normal Saline (Placebo Comparator): Ultrasound-guided suprainguinal fascia iliaca compartment block with 40mls normal saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: 0.5% Ropivacaine — Ultrasound-guided suprainguinal fascia iliaca compartment block with 40mls 0.5% ropivacaine.
  Other Names: Naropin
  Arms: 0.5% Ropivacaine
Drug: Normal saline — Ultrasound-guided suprainguinal fascia iliaca compartment block with 40mls normal saline.
  Arms: Normal Saline

SUMMARY:
Total hip replacement (THR) is a common and major surgical procedure performed in elderly patients with significant comorbidities. Optimizing a patient's anesthetic and analgesic modalities could play a significant role in minimizing the risk of adverse events in the perioperative period and potentially shorten time to discharge and recovery.

Establishing a safe and effective post-operative analgesic plan is of central importance to successful THR anesthesia care. The application of ultrasound visualization has improved the efficacy of the fascia iliaca compartment block (FICB). However, ultrasound-guided suprainguinal FICB has not yet been evaluated clinically in a large trial as a method of providing post-operative analgesia following THR.

The investigators hypothesize that by performing the suprainguinal fascia iliaca block with ultrasound, it will be possible to achieve superior and more reliable analgesia in the first 24 hours than without a block.

DETAILED DESCRIPTION:
The search for the optimal pain treatment strategies is a work in progress. As techniques and technology evolve so should our approach for the best analgesic regimen that would minimize unwanted side effects and potential risk and more importantly improve patient satisfaction.

The literature has supported the use of peripheral nerve blocks for analgesia as well as improved functional outcome after total knee arthroplasty. The addition of peripheral nerve blocks for THR has been more controversial, as the only effective nerve block, the posterior approach to the lumbar plexus, is an advanced regional technique with potential for serious complications. The application of ultrasound visualization has improved the efficacy of the infrainguinal fascia iliaca block. However, ultrasound guided suprainguinal fascia iliaca block has not yet been evaluated clinically in a large trial as a method of providing post-operative analgesia following primary hip arthroplasty.

The investigators hypothesize that by performing the suprainguinal fascia iliaca block with ultrasound, it will be possible to achieve superior and more reliable analgesia than that obtained using the landmark "2-pop" technique and the infrainguinal blocks.

The aim of this study is to assess whether the ultrasound guided suprainguinal fascia iliaca block can provide superior early postoperative analgesia in patients undergoing primary hip arthroplasty, and minimizing the pain immediately after the resolution of the spinal anesthetic.

The investigators propose to perform the first triple-blinded RCT examining the early analgesic efficacy of ultrasound-guided suprainguinal FICB after THR (lateral approach) under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75, ASA I-III scheduled to undergo unilateral total hip arthroplasty.

Exclusion Criteria:

* Patients not providing informed consent.
* Refusal of treatment plan.
* Pre-existing medical/neurological/hematologic conditions contraindicated for spinal anesthesia or peripheral nerve blocks.
* Revision total hip arthroplasty.
* Known allergy to any of the medications being used.
* History of drug or alcohol abuse.
* Patients with chronic pain on slow-release preparations of opioid in excess of 30mg of morphine equivalence per day.
* Patients with Rheumatoid Arthritis.
* Patients with psychiatric disorders.
* Patients with prior surgery in the inguinal region or inguinal hernia
* Patients unable or unwilling to use Patient Control Analgesia.
* Diabetic patients with diabetic neuropathy or those with impaired renal function (Creatinine >106).
* Patients with BMI >45.
* Patients with body weight <65kg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption at 24 hours after arrival in post-operative care unit | 24 hours
  Opioid consumption at 24 hours after arrival in PACU amongst the various treatment groups will be our primary outcome. Opioid usage for the first 24 hours will be simply determined from the patient-controlled analgesia data in addition to oral narcotics administered.

SECONDARY OUTCOMES:
Pain Scores | Every 4 hours after arrival in post-operative care unit for 24 hours
  Numerical Rating Scale (NRS-11) for pain will be used (0=no pain, 10=terrible pain) as the secondary outcome measure. The NRS score will be recorded on arrival to PACU and every 4 hours thereafter for 24 hours at rest and during mobilization by the treating ward nurse.
Respiratory Depression | Every 4 hours after arrival in post-operative care unit for 24 hours
  Respiratory rate will be recorded on arrival to PACU and every 4 hours thereafter for 24 hours. Respiratory depression will be defined as respiratory rate less than 10 breaths per minute.
Nausea | Every 4 hours after arrival in post-operative care unit for 24 hours
  Nausea will be recorded on arrival to PACU and every 4 hours thereafter for 24 hours.
  Nausea and Vomiting Scale:
  0 = No N & V
  1. = Mild N & V, no treatment required
  2. = Severe N & V, treatment required
  3. = Treatment effective
  4. = Treatment ineffective
Vomiting | Every 4 hours after arrival in post-operative care unit for 24 hours
  Vomiting will be recorded on arrival to PACU and every 4 hours thereafter for 24 hours.
  Nausea and Vomiting Scale:
  0 = No N & V
  1. = Mild N & V, no treatment required
  2. = Severe N & V, treatment required
  3. = Treatment effective
  4. = Treatment ineffective
Pruritus | Every 4 hours after arrival in post-operative care unit for 24 hours
  Pruritus will be recorded on arrival to PACU and every 4 hours thereafter for 24 hours.
  Pruritus Scale:
  0 = No pruritis
  1. = Mild pruritis, no treatment required
  2. = Severe pruritis, treatment required
  3. = Treatment effective
  4. = Treatment ineffective

CONTACTS AND LOCATIONS:
Locations (1):
- Holland Orthopedic and Arthritic Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Safa B, Trinh H, Lansdown A, McHardy PG, Gollish J, Kiss A, Kaustov L, Choi S. Ultrasound-guided suprainguinal fascia iliaca compartment block and early postoperative analgesia after total hip arthroplasty: a randomised controlled trial. Br J Anaesth. 2024 Jul;133(1):146-151. doi: 10.1016/j.bja.2024.04.019. Epub 2024 May 18. PMID 38762396